CLINICAL TRIAL: NCT00049218
Title: A Phase I-II Trial Using Dendritic Cells Transduced With An Adenoviral Vector Containing The p53 Gene To Immunize Patients With Extensive Stage Small Cell Lung Cancer After Standard Chemotherapy
Brief Title: Chemotherapy Followed By Vaccine Therapy in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13427; 0205-538 (Other: OBA)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine Administration (Experimental): • Phase I: Beginning 9 weeks after completion of chemotherapy, patients receive autologous dendritic cell-adenovirus p53 vaccine subcutaneously (SC) on days 1, 14, and 28. Patients without PD may undergo repeat leukapheresis on day 49. Patients receive vaccine SC again on days 56, 84, and 112 in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of autologous dendritic cell-adenovirus p53 vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  • Phase II: Patients receive autologous dendritic cell-adenovirus p53 vaccine at the MTD determined in phase I.
  Interventions: Biological: Autologous dendritic cell-adenovirus p53 vaccine; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Biological: Autologous dendritic cell-adenovirus p53 vaccine
Drug: Carboplatin
Drug: Etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Vaccines made from a gene-modified virus may make the body build an immune response to kill tumor cells. Combining vaccine therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of chemotherapy followed by adenovirus p53 vaccine therapy in treating patients who have extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of autologous dendritic cell-adenovirus p53 vaccine, administered after standard chemotherapy, in patients with extensive stage small cell lung cancer.
* Determine the toxicity of this regimen in these patients.
* Determine the development of an anti-p53-specific immune response in these patients after treatment with this regimen.
* Determine the tumor response rate, time to progression, and overall survival of patients treated with this regimen.
* Determine the frequency of anti-adenovirus immune responses in these patients after treatment with this regimen.

OUTLINE: This is a dose-escalation study of autologous dendritic cell-adenovirus p53 vaccine.

Patients undergo leukapheresis and dendritic cells are cultured. Adenovirus carrying p53 gene particles are added to the dendritic cells to make the vaccine. Leukapheresis is performed before chemotherapy or 8 weeks after the last dose of chemotherapy if the patient has already started chemotherapy.

Patients receive standard chemotherapy before receiving the vaccine. The recommended regimen is carboplatin IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients with progressive disease (PD) at 6 weeks after chemotherapy are removed from the study.

Patients are followed at day 140 and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 43-58 patients (3-18 for phase I and 40 for phase II) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed small cell lung cancer

  * Extensive stage disease
* Measurable disease
* No uncontrolled central nervous system (CNS) metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* Not specified

Hematopoietic

* White blood count (WBC) greater than 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hematocrit greater than 25%

Hepatic

* Bilirubin less than 2.0 mg/dL

Renal

* Creatinine less than 2.0 mg/dL

Immunologic

* HIV negative
* No serious ongoing infection
* No pre-existing immunodeficiency
* No known pre-existing autoimmune disorder

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* At least 4 weeks since prior steroids (before vaccination)
* No concurrent chronic steroids (during vaccination)

Radiotherapy

* At least 2 weeks since prior radiotherapy (before vaccination)

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-04; Primary Completion 2007-06 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Rate of Toxicity of the Ad-p53 DC Vaccine | 4 years
  To evaluate the toxicity of the Ad-p53 dendritic cell (DC) vaccine. While there is no expected toxicity from the Ad-p53 vaccine, there may be unforeseen adverse effects. Patients will be monitored for toxicity, particularly for evidence of autoimmunity. Complete blood counts (CBCs) to monitor for hematologic toxicity, serum creatinine to monitor for renal toxicity, liver function tests (LFTs) to monitor for hepatic toxicity, and a standard clinical toxicity will be performed every other week throughout the period of immunization. In addition, a medical history and physical examination will be performed on a monthly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Scott J. Antonia, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States